CLINICAL TRIAL: NCT04168164
Title: Aquatic Therapy in Patients With Adquired Brain Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, SAGRARIO PÉREZ DE LA CRUZ, Principal Investigator, Universidad de Almeria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UAlmeria
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Acquired Brain Injury
Keywords: aquatic therapy; balance; acquired brain injury.
MeSH Terms: conditions — Brain Injuries | interventions — Aquatic Therapy; Psychotherapy, Multiple

STUDY DESIGN:
Masking Description: This study was a randomized, single-blinded controlled trial. The participants were recruited from three brain injury associations and those who fulfilled the inclusion criteria were randomly assigned to three treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ai Chi (Experimental): Ai Chi aquatic therapy Dry land therapy
  Interventions: Other: aquatic therapy; Other: Dry land therapy; Other: Combined therapy

INTERVENTIONS:
Other: aquatic therapy — The exercises of Ai Chi were performed in a specific order, until completion of the total possible movements.
Other: Dry land therapy — sessions including exercises for gait, trunk mobility and exercises involving the upper and lower limbs
Other: Combined therapy — alternate sessions of therapy on dry land and aquatic therapy with Ai Chi

SUMMARY:
The aim of this study is to compare the relative effectiveness of three different treatment groups for improvements of postural control and for improvements of balance in these patients using aquatic therapy.

DETAILED DESCRIPTION:
Forty-five patients diagnosed with acquired brain injury, with over one year's evolution and independent gait over a distance of 10 meters, with our without the use of an orthopedic aid, were selected and randomized in 3 groups. Dry land therapy group (DT group), which received sessions including exercises for gait, trunk mobility and exercises involving the upper and lower limbs; Experimental group (EG group) , which received Ai Chi aquatic therapy; Combined group (DT+EG group), which received alternate sessions of therapy on dry land and aquatic therapy with Ai Chi.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of acquired brain injury traumatic or non-traumatic, with over one year's evolution
* the ability to walk independently over a distance of more than 10 meters, with or without an orthopedic aid
* scores on the Mini- Mental State Examination > 24

Exclusion Criteria:

* cardiovascular and/or respiratory problems, a previous history of neurological pathologiesand the presence of coadjuvants to the acquired brain injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 6 months
  The test consists of sitting, getting up, maintaining the standing position and changing positions, with a total of 14 items. The total possible score is 56 points, The scores on the Berg balance scale were classified as follows: high risk of falls (0-20), moderate risk (21-40) and low risk (> 41) with higher scores indicating that the person has better balance.
Five Times Sit-to-Stand test | 6 months
  The participants were seated with their arms crossed and they were asked to stand up and sit down five times as fast as possible

CONTACTS AND LOCATIONS:
Overall Officials: Sagrario Pérez- de la Cruz, Ph D, Principal Investigator — Universidad de Almeria
Locations (1):
- Sagrario, Almería, Spain